CLINICAL TRIAL: NCT03703167
Title: Phase Ib Trial With Dose Expansion of the Bruton"s Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, in Combination With Rituximab and Lenalidomide in Patients With Refractory/Recurrent Primary Central Nervous System Lymphoma (PCNSL) and Refractory/Recurrent Secondary Central Nervous System Lymphoma (SCNSL)
Brief Title: Ibrutinib With Rituximab and Lenalidomide for Patients With Recurrent/Refractory Primary or Secondary Central Nervous System Lymphoma (PCNSL/SCNSL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-432
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL); Secondary Central Nervous System Lymphoma (SCNSL)
Keywords: Ibrutinib; Rituximab; Lenalidomide; relapsed/refractory PCNSL; relapsed/refractory SCNSL; 18-432
MeSH Terms: conditions — Recurrence | interventions — ibrutinib; Lenalidomide; Rituximab

STUDY DESIGN:
Intervention Model Description: This is an open-label, phase Ib trial with dose expansion of the BTK inhibitor ibrutinib in combination with rituximab and lenalidomide.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ibrutinib in combination with rituximab and lenalidomide (Experimental): Ibrutinib will be given day 1-28; Lenalidomide will be given day 1-21; Rituximab will be given on day 1. Rituximab is given for 6 cycles; Lenalidomide is given for 12 cycles; Ibrutinib is continued until disease progression, intolerable toxicity or death.
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Oral ibrutinib will be given between days 1 and 28 of each 28-day cycle and will be continued daily after completion of rituximab and lenalidomide. The starting dose of ibrutinib is 560 mg/day (dose level 1) and (dose level 2 ibrutinib: 840 mg daily).
Drug: Lenalidomide — Oral lenalidomide will be given between days 1 and 21 of each 28-day cycle for a maximum of 12 cycles. The starting dose of lenalidomide is 10 mg/day (dose level 1 & 2) lenalidomide: 15 mg daily (dose level 3) and lenalidomide: 20 mg daily (dose level 4).
Drug: Rituximab — Intravenous rituximab (500mg/m2) will be given on day 1 of all cycles (+/- 3 days), for up to 6 cycles.

SUMMARY:
The investigator's want to find out if treatment with ibrutinib, rituximab, and lenalidomide are safe and better than the usual approach in patients with recurrent or refractory central nervous system lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to understand and be willing to sign a written informed consent document.
* Men and woman who are at least 18 years of age on the day of consenting to the study.
* Histologically documented PCNSL or histologically documented systemic diffuse large B-cell lymphoma (DLBCL).
* Patients must have relapsed/refractory PCNSL or relapsed/refractory SCNSL
* All patients need to have received at least one prior CNS directed therapy. There is no restriction on the number of recurrences.
* Patients with parenchymal lesions must have unequivocal evidence of disease progression on imaging (MRI of the brain or head CT) 21 days prior to study registration. For patients with leptomeningeal disease only, CSF cytology must document lymphoma cells and/or imaging findings consistent with CSF disease 21 days prior to study registration (at the discretion of the investigator).
* Participants must have an ECOG performance status of 0, 1, or 2.
* Participants must have adequate bone marrow and organ function shown by:

  * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
  * Platelets ≥ 75 x 10^9/L and no platelet transfusion within the past 21 days prior to study registration
  * Hemoglobin (Hgb) ≥ 8 g/dL and no red blood cell (RBC) transfusion within the past 21 days prior to study registration
  * International Normalized Ratio (INR) ≤ 1.5 and PTT (aPTT) ≤ 1.5 times the upper limit of normal
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal
  * Serum bilirubin ≤ 1.5 times the upper limit of normal; or total bilirubin ≤ 3 times the upper limit of normal with direct bilirubin within the normal range in patients with well documented Gilbert Syndrome.
  * Serum creatinine ≤ 2 times the upper limit of normal
  * Escalation: calculated creatinine clearance(CrCl) ≥ 60ml/min using the Cockcroft-Gault equation (Men: CrCl (min/ml) = (140-age) X (actual weight in kg) / 72 X serum creatinine (mg/dL); Women: CrCl (ml/min) = (140-age) X (actual weight in kg) X 0.85 / 72 X serum creatinine (mg/dL))
  * Extension: calculated creatinine clearance(CrCl) ≥30ml/min using the Cockcroft-Gault equation (Men: CrCl (min/ml) = (140-age) X (actual weight in kg) / 72 X serum creatinine (mg/dL); Women: CrCl (ml/min) = (140-age) X (actual weight in kg) X 0.85 / 72 X serum creatinine (mg/dL))
* Woman of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 30 days after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 3 months after the last dose.
* Female subjects of childbearing potential must have a negative plasma pregnancy test upon study entry. See section on Pregnancy and Reproduction.
* Patients must be able to tolerate MRI/CT scans.
* Patients must be able to tolerate lumbar puncture and/or Ommaya taps.
* Participants must have recovered to grade 1 toxicity from prior therapy.
* Participants should be able to submit up to 20 unstained formalin-fixed, paraffinembedded (FFPE) slides from the initial tissue diagnosis prior to study registration for confirmation of diagnosis and correlative studies
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.

NOTE: Prior autologous stem cell transplant as well as prior radiation to the CNS does NOT prevent patients from enrollment into the trial.

Exclusion Criteria:

* Patients with SCNSL actively receiving treatment for extra-CNS disease are excluded.
* Patient is concurrently using other approved or investigational antineoplastic agents.
* Patient has received chemotherapy, monoclonal antibodies or targeted anticancer therapy ≤ 4 weeks or 5 half-lives, whichever is shorter, or 6 weeks for nitrosourea or mitomycin-C prior to starting the study drug, or the patient has not recovered from the side effects of such therapy.
* Patient has received external beam radiation therapy to the CNS within 21 days of the first dose of the study drug.
* Patient requires more than 8 mg of dexamethasone daily or the equivalent
* Patient has an active concurrent malignancy requiring active therapy
* The patient has been treated with radio- or toxin-immunoconjugates within 70 days of the first dose of the study drug.
* Patient is allergic to components of the study drug.
* Patient is using warfarin or any other Coumadin-derivative anticoagulant or vitamin K antagonists. Patients must be off warfarin-derivative anticoagulants for at least seven days prior to starting the study drug. Low molecular weight heparin is allowed. Patients with congenital bleeding diathesis are excluded.
* Patient is taking a drug known to be a moderate and strong inhibitor or inducers of the P450 isoenzyme CYP3A. Participants must be off P450/CYP3A inhibitors and inducers for at least two weeks prior to starting the study drug.
* Patient is using systemic immunosuppressant therapy, including cyclosporine A, tacrolimus, sirolimus, and other such medications, or chronic administration of > 5 mg/day or prednisone or the equivalent. Participants must be off immunosuppressant therapy for at least 28 days prior to the first dose of the study drug.
* Patient has significant abnormalities on screening electrocardiogram (EKG) and active and significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, hypertension, valvular disease, pericarditis, or myocardial infarction within 6 months of screening,
* Patient has a known bleeding diathesis (e.g. von Willebrand"s disease) or hemophilia.
* Patient is known to have human immunodeficiency virus (HIV) infection.
* Patient is known to have a history of active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) as determined by serologic tests.
* Patient is known to have an uncontrolled active systemic infection.
* Patient underwent major systemic surgery ≤ 4 weeks prior to starting the trial treatment or who has not recovered from the side effects of such surgery, or who plan to have surgery within 2 weeks of the first dose of the study drug.
* Patient is unable to swallow capsules or has a disease or condition significantly affecting gastrointestinal function, such as malabsorption syndrome, resection of the stomach or small bowel, or complete bowel obstruction.
* Patient has poorly controlled diabetes mellitus with a glycosylated hemoglobin >8% or poorly controlled steroid-induced diabetes mellitus with a glycosylated hemoglobin of >8%. (for patients who received a short-term, high-dose dexamethasone treatment course prior to enrollment (<7 days), the HbA1c value can be rounded to the nearest whole number).
* Patient has a life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the investigator, could compromise the subject"s safety or put the study outcomes at undue risk.
* Women who are pregnant or nursing (lactating), where pregnancy is defined as a state of a female after conception until the termination of gestation, confirmed by a positive serum hCG laboratory test of > 5 mIU/mL (See section on Pregnancy and Reproduction)
* Patient has undergone prior allogenic stem cell transplant (autologous stem cell transplant is NOT an exclusion)
* The patient is unwell or unable to participate in all required study evaluations and procedures
* Known hypersensitivity to ibrutinib, thalidomide or lenalidomide
* Females who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2026-01-26 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) of ibrutinib | 1 year
  A standard 3+3 design will be employed. Four dose levels will be investigated. Patients will be treated in cohorts of size three to six and the dosage will be escalated if the clinical toxicity is acceptable. A dose limiting toxicity (DLT) is defined as in any of the following during cycle 1: any grade 4 hematologic toxicity, grade 3 febrile neutropenia and grade 3 thrombocytopenia associated with bleeding or any grade ≥3 non-hematologic toxicity that does not respond to supportive therapy and at least possibly related to treatment with ibrutinib. A minimum of 4 up to a maximum of 30 patients will be enrolled.

SECONDARY OUTCOMES:
progression free survival | 2 years
  Progression-free survival (PFS) is defined as the time from the date of treatment start to the date of the first documented PD or death due to any cause. If a patient is not known to have progressed or died at the date of the analysis cut-off or when he/she receives any further anti-cancer therapy, PFS is censored at the time of the last tumor assessment before the cutoff date and before the anti-cancer therapy date. PFS will be based on the investigator"s assessment of MRI, CSF studies and clinical presentation.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grommes, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Schaff LR, Piotrowski AF, Pentsova E, Gavrilovic IT, Lin A, Kaley TJ, Wongchai V, Emadi-Paramkouhi L, Madzsar J, Quinn L, Gonzalez A, Breakey L, Tang SS, Mendez JS, Malani R, Nolan C, Hatzoglou V, Young RJ, DeAngelis LM, Reiner AS, Panageas KS, Francis JH, Mellinghoff IK, Grommes C. Phase Ib study with expansion of ibrutinib, lenalidomide, and rituximab in patients with relapsed/refractory central nervous system lymphoma. Neuro Oncol. 2025 Sep 17;27(8):2107-2116. doi: 10.1093/neuonc/noaf104. PMID 40269592
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm